CLINICAL TRIAL: NCT00824980
Title: Combined Inhibition of Dipeptidyl Peptidase IV (DPIV/CD26) and Aminopeptidase N (APN/CD13) in the Treatment of Psoriasis - Phase II Single Center Study
Brief Title: Combined Inhibition of Dipeptidyl Peptidase IV (DPIV/CD26) and Aminopeptidase N (APN/CD13) in the Treatment of Psoriasis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Immune Technologies & Medicine GmbH (Industry)
Responsible Party: Curdin Conrad, M.D., Dermatologische Klinik, Gloriastrasse 31, USZ, CH-8091 Zürich
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IMTM_IP10.C8_II/1
Record Dates: First submitted 2009-01-16; First posted 2009-01-19 (Estimated); Last update posted 2009-01-19 (Estimated); Status verified 2009-01

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- IP10.C8 Gel (Experimental)
  Interventions: Drug: IP10.C8
- Placebo Gel (Placebo Comparator)
  Interventions: Drug: IP10.C8

INTERVENTIONS:
Drug: IP10.C8 — IP10.C8 Gel 1%

SUMMARY:
The major objective of this study is to evaluate the therapeutic effect of a topical treatment simultaneously inhibiting Dipeptidyl Peptidase IV and Aminopeptidase N (IMTM #IP10.C8) in patients with mild to moderate psoriasis of the skin

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years of age at pre-study and
2. Diagnosis of plaque type psoriasis at least 3 month prior to enrolment
3. Mild to moderate plaque type psoriasis with at least 2 plaques of approximately 15cm2 for which topical treatment is indicated
4. Patients must be able to give written informed consent before any trial-specific procedures are performed (see Section 12.2

Exclusion Criteria:

1. Other type of psoriasis (e.g. erythrodermic, guttate or pustular) at enrolment
2. Drug induced psoriasis at enrolment (e.g. lithium)
3. Pregnant or lactating women, patients (men or women) planning a pregnancy during the duration of the study
4. Systemic therapy affecting PASI or phototherapy for a period of 4 weeks prior to enrolment
5. Topical therapy affecting PASI for a period of 2 weeks prior to enrolment
6. Treatment with biologic agents affecting PASI for a period of 3 months prior to enrolment
7. Systemic treatment with immunosuppressive agents (e.g. methotrexate, cyclosporin) or treatment with lithium, anti-malaria medication, or intramuscular gold application for a period of 4 weeks prior to enrolment
8. Having a history of or an ongoing uncontrolled serious or recurring bacterial, viral, fungal, or atypical mycobacterial infection
9. Having a severe medical condition that, in the judgment of the investigator, would jeopardize in any way the subject's safety following exposure to study drug
10. Having the presence or history of malignancy, including lymphoproliferative disorders. Subjects with a history of fully resolved basal or squamous cell skin cancer may be enrolled

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2009-01; Primary Completion 2009-09 (Estimated); Study Completion 2009-09 (Estimated)

PRIMARY OUTCOMES:
Psoriasis Area and Severity Index | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Lars E French, Prof., Principal Investigator — University Hospital Zurich Department of Dermatology / Gloriastrasse 31
Locations (1):
- University Hospital Zurich, Zurich, Switzerland